CLINICAL TRIAL: NCT07282080
Title: Discover Better Body Composition With Green Light!
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Efforia, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 43172
Record Dates: First submitted 2025-12-05; First posted 2025-12-15 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Body Composition

STUDY DESIGN:
Intervention Model Description: Single Arm observational where participants act as their own control
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single arm where participants act as their own control (Experimental): Single arm where participants act as their own control
  Interventions: Device: EmeraldLED

INTERVENTIONS:
Device: EmeraldLED — This device is a customizable, multi-wavelength therapeutic system designed for individualized cosmetic treatments. It features an easy-to-use interface with preprogrammed treatment categories, a wide pulsing frequency range from 1 to 15,000 Hz, and independent wavelength control for precise protocol tailoring. The system delivers five wavelengths-450 nm, 525 nm, 650 nm, 810 nm, and 980 nm-with an output power of 3,325 W and irradiance up to 119 mW/cm².
  The green light EmeraldLED therapy provided in this study is set at 525 nm.

SUMMARY:
Investigation into Green Light Therapy study using EmeraldLED for 15-minute sessions, twice a week, to support positive changes in body composition.

DETAILED DESCRIPTION:
This remotely administered decentralized trial is designed to rigorously explore the efficacy of green light therapy in influencing body composition and overall well-being. Under the leadership of Ryan, CEO of beem® Light Sauna, this study leverages the expansive network of over 50 wellness franchise locations across the United States, along with 30 years of fitness and wellness industry experience, to investigate the science-backed potential of green light therapy. Amidst the widespread speculation and anecdotal evidence circulating on social media, investigators seek to provide concrete, personalized data to participants, thereby empowering them with the knowledge to make informed decisions about their health and wellness strategies.

The core objective of this online study is to empower participants by providing a detailed analysis of how exposure to green light impacts their weight management journey and overall sense of well-being. By participating in this study, individuals will receive tailored feedback on their body composition changes and psychological well-being, offering a unique opportunity to understand the potential benefits of green light therapy on a personal level.

Participants in this remotely conducted trial will engage with state-of-the-art green light therapy sessions from the comfort of their chosen environment, ensuring a broad and inclusive participant base without geographic limitations. This approach not only facilitates a more diverse data set but also aligns with our commitment to making health innovations accessible to a wider audience.

The significance of this study cannot be overstated, as it aims to demystify the claims surrounding green light therapy and its effects on weight management and mental health. By contributing to this pioneering research, participants will be at the forefront of a potential paradigm shift in the approach to wellness and body composition optimization. While acknowledging the limitations of this study and the need for further extensive trials, the insights gained here will be invaluable in guiding future health innovations and strategies, marking a significant step towards a healthier, more informed society.

ELIGIBILITY:
Inclusion Criteria:

* Can read and understand English.
* US resident.
* Willing and able to follow the requirements of the protocol.

Exclusion Criteria:

-individuals with eye conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Body Image and Self-Perception Survey | Change from baseline (Day 1-3) in body image and self-perception at 4 weeks after the start of the intervention (Day 27-33)
  This survey aims to understand an individual's perception of their body, attractiveness, and physical functionality. It contains multiple-choice questions with five options ranging from 'Strongly Disagree' to 'Strongly Agree'. The questions are divided into three categories: Body Satisfaction, Attractiveness Evaluation, and Physical Functionality Awareness.
Body Composition Measurement Form | Change from baseline (Day 1-3) in body composition measurements at 4 weeks after the start of the intervention (Day 27-33)
  The Body Composition Measurement Form is specifically crafted to accurately track changes in body measurements relevant to individuals engaged in weight loss or bodybuilding. This form allows for the consistent recording of key physical metrics across various body parts, facilitating the evaluation of fitness progress. By using this form, individuals can obtain a clear picture of the physical changes resulting from their exercise routines and nutritional choices. Each measurement is to be recorded in centimeters to maintain uniformity and precision.
Quality of Life and Health Survey | Change from baseline (Day 1-3) in quality of life and health perceptions at 4 weeks after the start of the intervention (Day 27-33)
  This survey asks about your feelings towards your quality of life, health, and various areas of your life. It covers your experiences and feelings in the past four weeks. Please choose the answer that appears most appropriate.

CONTACTS AND LOCATIONS:
Locations (1):
- Efforia, New York, New York, United States

REFERENCES:
- See also: Additional information and join instructions on Efforia — https://app.efforia.com/wp-admin/admin.php?page=llms-course-builder&course_id=43167